CLINICAL TRIAL: NCT05928663
Title: The Effect on Puncture of the Use of Double Gloves in Orthopedic Surgery
Brief Title: The Effect of Using Double Gloves on Perforation in Orthopedic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Hülya Kızıl Toğaç, Principal Investigator, Celal Bayar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MCBÜ-HulyaKizilTogac
Record Dates: First submitted 2023-06-14; First posted 2023-07-03 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Puncture; Surgical Gloves; Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Gloves, Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- double surgical gloves (Experimental)
  Interventions: Other: double surgical gloves
- single surgical gloves (Other)
  Interventions: Other: single surgical gloves

INTERVENTIONS:
Other: double surgical gloves — In the intervention group, the surgical team members wore brown colored ENCORE® Latex Micro as the inner glove, while white MEDI-GRIP® Latex Standard was used as the outer glove
  Arms: double surgical gloves
Other: single surgical gloves — MEDI-GRIP® Latex Standard surgical gloves were included in the study as a single layer sterile surgical glove in the control group
  Arms: single surgical gloves

SUMMARY:
Aim: This study aimed to investigate the effect of using double gloves on perforation in orthopedic surgery.

Materials and Method: The randomized controlled experimental study was conducted between 30.11.2021 and 31.03.2022 in the Orthopedics and Traumatology operating room of a university hospital in western Turkey. The gloves used in the surgery were randomly divided into two groups (intervention: double glove group = 780 gloves, control: single glove group = 390). The presence of holes was checked by performing a water tightness test with the EN455-1 method on all gloves collected after the surgery by the researcher. Data were evaluated with descriptive statistics, Chi-square Test, Fisher Exact Test, and linear model regression analysis (GLM for the Binomial Family Regression). Statistical significance was accepted as 0.05.

DETAILED DESCRIPTION:
The sample size of the study was calculated based on the work of Makama et al. In the study, the perforation rate of the single glove was 15.2% and the perforation rate of the second glove in the double glove was determined as 1.17%. Considering these values, the number of gloves to be included in the intervention and control groups (in the single and double glove groups) was calculated as 249, with a 99% confidence interval (α=0.001) and 99% power in the NCSS PASS program. The total number of gloves planned to be evaluated in the intervention (double glove group, 249x2=498) and control (single glove group, 249) groups was determined as 747. The study included a total of 1170 gloves, with 780 gloves in the intervention group and 390 gloves in the control group. The allocation of gloves to the groups was determined using block randomization. The block size of 4 was selected, and all possible permutations of allocation within the block were computed. Blocks were then randomly selected to indicate the allocation of gloves to the intervention or control group.

Data Collection Tools

Patient and Surgery Information Form: In this form, which was created by examining the researches on glove perforations, there are 13 questions consisting of information about the patient, information about the surgical procedure and information about the surgical team.

Gloves Information Form: In this form, which was prepared by examining the literature, there are 16 questions such as the type of glove collected after the surgery, the team member using the glove, the dominant hand of the person using the glove, the duration of experience, the use of cement in the surgery, the time and reasons for replacing the gloves, the perforation conditions, the areas where the perforations are located Interventions Before the research, the necessary approval (Reference number: 20.05.2020/20.478.486) was obtained from the university clinical ethics committee, and the research was performed according to the principles of the Helsinki Declaration. Orthopedic surgeries other than soft tissue surgeries were included in the study.

When the patient was admitted to the operating room, the section containing the patient's information was filled out by using the patient file. On the same form, it was filled in the section containing the information about the surgical team and recorded in the form. In the intervention group, the surgical team members wore brown colored ENCORE® Latex Micro as the inner glove, while white MEDI-GRIP® Latex Standard was used as the outer glove. In the control group, only MEDI-GRIP® Latex Standard gloves were worn. All information about the gloves used in the surgery was recorded in the forms prepared by the researcher. In these forms, the team member who used the gloves, if the gloves were changed, the reason for the change and the time of replacement were stated. Making the surgical incision was defined as the beginning of the operation and the end of the operation when the incision was closed and all surgical instruments were removed from the patient. The time between the beginning and the end of the surgery in minutes was recorded on the form. The number of single and double gloves used during the surgery, the duration of the surgery and the cutting and piercing rotary devices and tools that may affect the perforations were also recorded on the forms. During the operation, the members of the surgical team were constantly monitored by the researcher. In cases where glove change was made, the reason and time of glove change were recorded by the researcher. The gloves used were placed in boxes with barcodes before hand.

All gloves collected after the surgery were tested by the researcher by standardized water leak method EN 455-1. In this method, which was applied to determine the perforation status in the gloves, 1000±50 ml of tap water was filled into the gloves. The temperature of the water was between 15-35°C. Gloves filled with water were observed for two minutes. The area where the water leak occurred was marked on the form and recorded. All fingers were lettered, starting with the little finger of the left hand, in order to more easily register the perforation areas in the gloves (left pinky: a, right pinky: j, left back: k, right back: l, left palm: m, and right palm: n). The perforations detected during the water tightness control were recorded in this order. The same test was applied to the gloves that were opened and not used for control purposes at the beginning of each operation. In the study, double gloves were worn in 55 operations in the intervention group, while single gloves were worn in 57 operations in the control group. Gloves of the same brand, which were opened on the operating table but never used, were checked for each operation. No perforations were detected total of 334 in these gloves that 220 (inner gloves 55x2=110; outer gloves 55x2=110) in the intervention group and 114 (57x2=114) in the control group. Although the number of people in the surgical team during the operation was not standard, there was definitely a surgeon and a nurse in the team. The water leak test applied to collect the gloves used after the surgery and to detect the perforations was performed by the same researcher. However, the same person who was a nurse among the surgical team members during the water leak test of all gloves was present as an observer at the time of the test.

ELIGIBILITY:
Inclusion Criteria:

* In the intervention group, ENCORE® Latex Micro was used as the inner glove and MEDI-GRIP® Latex Standard was used as the outer glove
* MEDI-GRIP® Latex Standard gloves were used in the control group.

Exclusion Criteria:

* Gloves that were removed before the operation starts in cases where the surgical team member's glove is torn or contaminated for any reason.
* Gloves worn by the surgical team member after changing gloves for any reason.
* Gloves worn by the replacement person in cases where the surgical team members leave their place to another team member for any reason.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1170 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Investigation of Perforations Presence of Gloves by Groups | immediately after surgery
  Whether there is a puncture (perforation) or not in intervention and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Hakan BAYDUR, Assoc. Prof., Study Chair — Manisa Celal Bayar University, Faculty of Health Sciences
Locations (1):
- Manisa Celal Bayar University Faculty of Health Sciences, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bashaw MA, Keister KJ. Perioperative Strategies for Surgical Site Infection Prevention. AORN J. 2019 Jan;109(1):68-78. doi: 10.1002/aorn.12451. PMID 30592511
- [Background] Bekele A, Makonnen N, Tesfaye L, Taye M. Incidence and patterns of surgical glove perforations: experience from Addis Ababa, Ethiopia. BMC Surg. 2017 Mar 20;17(1):26. doi: 10.1186/s12893-017-0228-8. PMID 28320370
- [Background] de Barros MPM, Godoi TTF, Ferretti Filho M, Fernandes HJA, Dos Reis FB. Surgical Gloves in Orthopedic Trauma Procedures: How Many Lose Their Integrity? Rev Bras Ortop (Sao Paulo). 2021 Jun;56(3):379-383. doi: 10.1055/s-0040-1722591. Epub 2021 Jul 1. PMID 34239206
- [Background] Egeler K, Stephenson N, Stanke N. Glove perforation rate with orthopedic gloving versus double gloving technique in tibial plateau leveling osteotomy: A randomized trial. Can Vet J. 2016 Nov;57(11):1156-1160. PMID 27807378
- [Background] Ellis H. Surgical gloves. J Perioper Pract. 2010 Jun;20(6):219-20. doi: 10.1177/175045891002000606. PMID 20586363
- [Background] Gaines S, Luo JN, Gilbert J, Zaborina O, Alverdy JC. Optimum Operating Room Environment for the Prevention of Surgical Site Infections. Surg Infect (Larchmt). 2017 May/Jun;18(4):503-507. doi: 10.1089/sur.2017.020. Epub 2017 Apr 12. PMID 28402706
- [Background] Goldman AH, Haug E, Owen JR, Wayne JS, Golladay GJ. High Risk of Surgical Glove Perforation From Surgical Rotatory Instruments. Clin Orthop Relat Res. 2016 Nov;474(11):2513-2517. doi: 10.1007/s11999-016-4948-3. Epub 2016 Jun 23. PMID 27339122
- [Background] Jid LQ, Ping MW, Chung WY, Leung WY. Visible glove perforation in total knee arthroplasty. J Orthop Surg (Hong Kong). 2017 Jan;25(1):2309499017695610. doi: 10.1177/2309499017695610. PMID 28228047
- [Background] Lakomkin N, Cruz AI Jr, Fabricant PD, Georgiadis AG, Lawrence JTR. Glove Perforation in Orthopaedics: Probability of Tearing Gloves During High-Risk Events in Trauma Surgery. J Orthop Trauma. 2018 Sep;32(9):474-479. doi: 10.1097/BOT.0000000000001233. PMID 29889823
- [Background] Lathan SR. Rubber gloves redux. Proc (Bayl Univ Med Cent). 2011 Oct;24(4):324. doi: 10.1080/08998280.2011.11928750. No abstract available. PMID 22046069
- [Background] Lee SW, Cho MR, Lee HH, Choi WK, Lee JH. Perforation of Surgical Gloves during Lower Extremity Fracture Surgery and Hip Joint Replacement Surgery. Hip Pelvis. 2015 Mar;27(1):17-22. doi: 10.5371/hp.2015.27.1.17. Epub 2015 Mar 31. PMID 27536597
- [Background] Lee SY. What Role Does a Colored Under Glove Have in Detecting Glove Perforation in Foot and Ankle Procedures? Clin Orthop Relat Res. 2022 Dec 1;480(12):2327-2334. doi: 10.1097/CORR.0000000000002268. Epub 2022 Jun 2. PMID 35695671
- [Background] Lindsey RW. CORR Insights(R): High Risk of Surgical Glove Perforation From Surgical Rotatory Instruments. Clin Orthop Relat Res. 2016 Nov;474(11):2518-2521. doi: 10.1007/s11999-016-5004-z. Epub 2016 Aug 10. No abstract available. PMID 27511200
- [Background] Link T. Guideline Implementation: Sterile Technique. AORN J. 2019 Oct;110(4):415-425. doi: 10.1002/aorn.12803. PMID 31560430
- [Background] Makama JG, Okeme IM, Makama EJ, Ameh EA. Glove Perforation Rate in Surgery: A Randomized, Controlled Study To Evaluate the Efficacy of Double Gloving. Surg Infect (Larchmt). 2016 Aug;17(4):436-42. doi: 10.1089/sur.2015.165. Epub 2016 Mar 16. PMID 26981792
- [Background] O'Hara LM, Thom KA, Preas MA. Update to the Centers for Disease Control and Prevention and the Healthcare Infection Control Practices Advisory Committee Guideline for the Prevention of Surgical Site Infection (2017): A summary, review, and strategies for implementation. Am J Infect Control. 2018 Jun;46(6):602-609. doi: 10.1016/j.ajic.2018.01.018. Epub 2018 Mar 7. PMID 29525367
- [Background] Osborne MP. William Stewart Halsted: his life and contributions to surgery. Lancet Oncol. 2007 Mar;8(3):256-65. doi: 10.1016/S1470-2045(07)70076-1. PMID 17329196
- [Background] Salassa TE, Swiontkowski MF. Surgical attire and the operating room: role in infection prevention. J Bone Joint Surg Am. 2014 Sep 3;96(17):1485-92. doi: 10.2106/JBJS.M.01133. PMID 25187588
- [Background] Schlich T. Why were surgical gloves not used earlier? Lancet. 2015 Sep 26;386(10000):1234-5. doi: 10.1016/S0140-6736(15)00271-8. No abstract available. PMID 26460651
- [Background] Spruce L. Back to Basics: Sterile Technique. AORN J. 2017 May;105(5):478-487. doi: 10.1016/j.aorn.2017.02.014. PMID 28454613
- [Background] Tao LX, Basnet DK. Study of Glove Perforation during Hip Replacement Arthroplasty: Its Frequency, Location, and Timing. Int Sch Res Notices. 2014 Oct 29;2014:129561. doi: 10.1155/2014/129561. eCollection 2014. PMID 27350965
- [Background] Thomson I, Krysa N, McGuire A, Mann S. Recognition of intraoperative surgical glove perforation: a comparison by surgical role and level of training. Can J Surg. 2022 Feb 8;65(1):E82-E88. doi: 10.1503/cjs.016720. Print 2022 Jan-Feb. PMID 35135784
- [Background] Tlili MA, Belgacem A, Sridi H, Akouri M, Aouicha W, Soussi S, Dabbebi F, Ben Dhiab M. Evaluation of surgical glove integrity and factors associated with glove defect. Am J Infect Control. 2018 Jan;46(1):30-33. doi: 10.1016/j.ajic.2017.07.016. Epub 2017 Sep 20. PMID 28893444
- [Background] Wacholder S. Binomial regression in GLIM: estimating risk ratios and risk differences. Am J Epidemiol. 1986 Jan;123(1):174-84. doi: 10.1093/oxfordjournals.aje.a114212. PMID 3509965
- [Background] Zaatreh S, Enz A, Klinder A, Konig T, Mittelmeier L, Kundt G, Mittelmeier W. Prospective data collection and analysis of perforations and tears of latex surgical gloves during primary endoprosthetic surgeries. GMS Hyg Infect Control. 2016 Dec 20;11:Doc25. doi: 10.3205/dgkh000285. eCollection 2016. PMID 28066701
- [Background] Zhang Z, Gao X, Ruan X, Zheng B. Effectiveness of double-gloving method on prevention of surgical glove perforations and blood contamination: A systematic review and meta-analysis. J Adv Nurs. 2021 Sep;77(9):3630-3643. doi: 10.1111/jan.14824. Epub 2021 Mar 17. PMID 33733484
- [Background] AORN. Guideline at a Glance: Sharps Safety. AORN J. 2017 Jul;106(1):87-89. doi: 10.1016/S0001-2092(17)30527-6. No abstract available. PMID 28662791

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT05928663/Prot_SAP_000.pdf